CLINICAL TRIAL: NCT07275177
Title: Effect of Vitamin D Supplementation on Strength and Muscle Gain in Older Adults With Obesity in Miahuatlán de Porfirio Díaz, in Period 2023-2024
Brief Title: Effect of Vitamin D on Body Composition and Functionality of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma Benito Juárez de Oaxaca (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Carlos Valencia Santiago, Principal Investigator, Universidad Autónoma Benito Juárez de Oaxaca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESV/CIUU/290923
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Disorder); Obesity; Sarcopenia; Sarcopenia in Elderly; Sarcopenic Obesity; Vitamin D Deficiency; Vitamin D 25-Hydroxylase Deficiency; Muscle Strengh; Muscle Mass; Aging; Older Adults (65 Years and Older); Functional Decline; Age-Related Loss of Skeletal Muscle Mass; Muscle Weakness
Keywords: Sarcopenic Obesity; Obesity; Sarcopenia; Vitamin D deficiency; Muscle Weakness; Functional Decline; Aging; Older Adults
MeSH Terms: conditions — Obesity; Sarcopenia; Vitamin D Deficiency; Vitamin D Hydroxylation-Deficient Rickets, Type 1B; Muscle Weakness | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups. The intervention group received daily oral vitamin D3 (10,000 IU/day) for 12 weeks. The placebo group received a daily oral placebo capsule identical in appearance. All participants completed identical baseline and post-intervention assessments, including anthropometry, body composition, muscle strength, physical performance (SPPB), dietary intake, and serum 25(OH)D levels.
Who Masked: Participant
Masking Description: Participants were blinded to group assignment. Vitamin D3 capsules and placebo capsules were identical in size, color, and appearance. Investigators administering the supplementation and collecting outcomes were aware of allocation, but participants did not know whether they were receiving vitamin D or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplementation (Cholecalciferol) (Experimental): Participants receive oral vitamin D3 (cholecalciferol) at a dose of 10,000 IU per day for 12 weeks, in addition to their usual medical care. All participants undergo baseline and post-intervention assessments of muscle strength, muscle mass, functional performance, body composition, dietary intake, and serum 25(OH)D levels.
  Interventions: Dietary Supplement: Vitamin D
- Placebo capsule (Placebo Comparator): Daily oral placebo capsules for 12 weeks. Placebo capsules match the vitamin D capsules in size, shape, and appearance but contain inactive ingredients only.
  Interventions: Dietary Supplement: Vitamin D placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants receive oral vitamin D3 (cholecalciferol) at a dose of 10,000 IU per day for 12 weeks, in addition to their usual medical care. All participants undergo baseline and post-intervention assessments of muscle strength, muscle mass, functional performance, body composition, dietary intake, and serum 25(OH)D levels.
  Arms: Vitamin D supplementation (Cholecalciferol)
Dietary Supplement: Vitamin D placebo — Daily oral placebo capsules for 12 weeks. Placebo capsules match the vitamin D capsules in size, shape, and appearance but contain inactive ingredients only
  Arms: Placebo capsule

SUMMARY:
Older adults with obesity often experience a gradual loss of muscle mass and muscle strength, a condition sometimes described as sarcopenic obesity. This combination increases the risk of falls, disability, functional decline, and metabolic complications. Low levels of vitamin D are common in older adults and may contribute to reduced muscle function and poorer physical performance.

This study is designed to evaluate whether taking 10,000 International Units (IU) per day of vitamin D3 for 12 weeks can improve muscle strength and muscle mass in older adults with obesity living in southern Mexico. The study will also examine whether vitamin D3 supplementation influences body composition, physical performance, and serum levels of 25-hydroxyvitamin D.

Participants will complete assessments at the beginning and at the end of the 12-week period. These assessments include measurements of muscle strength, skeletal muscle mass, body fat percentage, and indicators of physical performance such as the Short Physical Performance Battery (SPPB). Additional measures of body composition and anthropometry, such as body mass index, waist circumference, and related indices, will also be recorded. Blood samples will be analyzed to determine vitamin D status.

All participants will receive daily oral vitamin D3 (cholecalciferol) throughout the 12-week intervention. The goal of the study is to understand whether improving vitamin D status can have a positive effect on muscle health and physical function in older adults with obesity.

The results from this research may help guide future strategies to prevent or reduce functional decline related to low muscle mass in older adults with obesity, particularly in rural regions of Mexico where vitamin D deficiency is common.

DETAILED DESCRIPTION:
This randomized controlled study investigated the effects of vitamin D3 supplementation on muscle strength, body composition, and functional performance in older adults with obesity. Vitamin D deficiency is highly prevalent in this population and has been associated with reduced skeletal muscle mass, decreased physical performance, increased fat accumulation, and progression toward frailty. Improving vitamin D status may contribute to better musculoskeletal health and improved physical function.

Participants received 10,000 International Units (IU) per day of vitamin D3 for a total period of 12 weeks. All assessments were conducted at baseline and at week 12. Handgrip strength was measured using a Jamar hand dynamometer as an indicator of muscle strength. Skeletal muscle mass, body fat percentage, visceral fat index, metabolic age, and related measures were obtained via Bioelectrical Impedance Analysis (BIA). Anthropometric variables including weight, body mass index (BMI), waist circumference, abdominal volume index (AVI), and body adiposity index (BAI) were also recorded.

Functional status was assessed using the Short Physical Performance Battery (SPPB), a validated tool consisting of balance, gait speed, and chair stand tests. The SPPB ranges from 0 to 12 points, with higher scores indicating better physical performance.

Serum concentrations of 25-hydroxyvitamin D [25(OH)D] were evaluated using standardized laboratory techniques to determine changes in vitamin D status associated with supplementation.

This study seeks to clarify whether vitamin D3 supplementation can improve muscle strength, muscle mass, functional performance, and body composition among older adults with obesity, and to better understand the role of vitamin D in age-related musculoskeletal decline.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older.
* Diagnosis of obesity (BMI ≥ 30 kg/m²).
* Patients attending the outpatient clinic of IMSS No. 24 in Miahuatlán de Porfirio Díaz, Oaxaca.
* Able to perform physical and functional tests (handgrip, SPPB).
* Capable of providing informed consent.
* Willing to comply with the intervention and attend baseline and 12-week evaluations.

Exclusion Criteria:

* Known diagnosis of hypercalcemia or disorders of calcium metabolism.
* Current use of high-dose vitamin D supplementation or medications affecting vitamin D metabolism.
* Severe renal or hepatic disease.
* Active cancer treatment.
* Neurological or musculoskeletal conditions that impair mobility or functional testing (e.g., recent fractures, severe osteoarthritis, stroke with major disability).
* Cognitive impairment preventing the understanding of instructions or informed consent.
* Any medical condition that, in the judgment of investigators, would interfere with participation or pose additional risk.
* Participation in another clinical trial during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Handgrip strehgth (kg) | Baseline and 12 weeks
  Muscle strength will be measured using a handheld dynamometer following standardized procedures. The highest value from two attempts per hand will be used. Results reported in kilograms (kg). Higher values indicate greater muscle strength.
Skeletal muscle mass | Baseline and 12 weeks
  Skeletal Muscle mass assessed by Bioelectrical Impedance Analysis (BIA). Results reported in kilograms (kg)

SECONDARY OUTCOMES:
Body Fat percentage | Baseline and 12 weeks
  Total body fat percentage measured using bioelectrical impedance analysis (BIA). The results will be expressed as a percentage (%)
Visceral Fat Index | Baseline and 12 weeks
  Visceral fat index obtained through Bioelectrical Impedance Analysis (BIA). The results will be expressed in index units
Body Adiposity Index (BAI) | Baseline and 12 weeks
  Body Adiposity Index calculated from hip circumference and height. The results will be expressed in index units
Short physical Performance Battery (SPPB) Score | Baseline and 12 weeks
  Functional performance assessed using the SPPB, wich includes balance tests, gait speed, and chair stands.
Serum 25-Hydroxyvitamin D Levels | Baseline and 12 weeks
  Serum levels of 25-hydroxyvitamin D [25(OH)D], measured in nanograms per mililiter (ng/mL)
SPPB Score | Baseline and 12 weeks
  Short Physical Performance Battery (SPPB) score, ranging from 0 (worst performance) to 12 (best performance). Higher scores indicate better physical function.
Weight | baseline and 12 weeks
  Body weight measured in kilograms (kg)
Body Mass Index (BMI) | Baseline and 12 weeks
  Body Mass Index (BMI) calculated as weight (kg) divided by height squared (m2). The results will be expressed in kg/m2
Waist circumference | Baseline and 12 weeks
  Waist circumference measured in centimeters (cm)
Metabolic Age | Baseline and 12 weeks
  Metabolic Age estimated by BIA based on body composition paremeters. The results will be expressed in years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Valencia Santiago, Doctor, Principal Investigator — Universidad Autónoma Benito Juárez de Oaxaca
Locations (1):
- Instituto Mexicano del Seguro Social - Unidad de Medicina Familiar 24, Miahuatlán de Porfirio Díaz, Oaxaca, México, Miahuatlán de Porfirio Díaz, Oaxaca, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study was conducted within a clinical care setting of IMSS and contains protected health information. Data are restricted by institutional and ethical regulations.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT07275177/Prot_ICF_000.pdf